CLINICAL TRIAL: NCT04530916
Title: Antihypertensive and Vascular-Protective Effects of Wild Blueberries in Middle-Aged/Older Men and Postmenopausal Women.
Brief Title: Wild Blueberries and Cardiovascular Health in Middle-aged/Older Men and Postmenopausal Women
Acronym: WB2020
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: Wild Blueberry Association of North America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1775
Record Dates: First submitted 2020-01-27; First posted 2020-08-28 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Hypertension; Aging; Endothelial Dysfunction; Men
Keywords: Cardiovascular Disease; Blueberries; Hypertension; Vascular Dysfunction; Atherosclerosis; Aging
MeSH Terms: conditions — Hypertension; Multiple Endocrine Neoplasia Type 1; Cardiovascular Diseases; Atherosclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blueberry (Experimental): 22 g blueberry powder per day
  Interventions: Dietary Supplement: Blueberry Powder
- Control (Placebo Comparator): 22 g placebo control powder per day
  Interventions: Dietary Supplement: Placebo Powder

INTERVENTIONS:
Dietary Supplement: Blueberry Powder — 22 g/day wild blueberry powder
  Arms: Blueberry
Dietary Supplement: Placebo Powder — 22 g/day placebo powder
  Arms: Control

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of morbidity and mortality worldwide. Aging is the primary risk factor for CVD, in large part due to adverse modifications to the arteries. These modifications include vascular endothelial dysfunction and arterial stiffness. Vascular endothelial dysfunction is an initiating step in atherosclerosis, and is primarily caused by reduced nitric oxide (NO) bioavailability secondary to excessive superoxide-driven oxidative stress and inflammation. Endothelial dysfunction leads to arterial stiffness and the development of hypertension (HTN) which further increases CVD. Greater than 2/3 of the US population has elevated blood pressure or stage 1-HTN. As such, interventions that improve vascular endothelial dysfunction by increasing NO bioavailability and mitigating excessive oxidative stress and inflammation are needed. Blueberries are rich in bioactive compounds including flavonoids, phenolic acids, and pterostilbene. These compounds and their metabolites have been shown to attenuate oxidative stress and inflammation. The primary goal of this study is to assess the efficacy of blueberries to improve reduce blood pressure and improve vascular endothelial dysfunction and arterial stiffness in middle-aged/older men with elevated blood pressure or stage 1-HTN.

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women
* Aged 45-70 years
* Elevated blood pressure or stage 1-Hypertension
* Ability to provide informed consent

Exclusion Criteria:

* Have had a menstrual cycle within the past year
* Blood Pressure < 120 (systolic BP) or ≥ 140/90 mm Hg
* Reactive hyperemia index > 3.00%
* Taking > 1 antihypertensive medication, taking 1 antihypertensive medication more than 1 time per day, and/or taking the antihypertensive medication for < 3 months
* Diagnosed cancer, cardiovascular disease, diabetes, or gastrointestinal, kidney, liver, lung, and/or pancreatic disease
* Triglycerides > 350 mg/dL, low-density lipoprotein cholesterol (LDL-C) ≥ 190 mg/dL, hemoglobin A1c ≥ 6.5%, and/or taking a lipid-lowering or glucose-lowering medication
* Testosterone or estrogen replacement therapy use 6 months prior to study start
* Weight change ≥ 3 kg in the past 3 months, actively trying to lose weight, or unwilling to remain weight stable throughout the study
* Current smokers or history of smoking in the past 12 months
* Binge and/or heavy drinker (>3 drinks on any given occasion and/or >7 drinks/week for women, and >4 drinks on any given occasion and/or >14 drinks/week for men)
* Body mass index < 18.5 or > 40 kg/m2
* Antibiotic therapy within past two months
* Allergies or contraindication to study treatments or procedures

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 58 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Reactive hyperemia index | Baseline to 12 Weeks
  Endothelial function assessed as reactive hyperemia index using peripheral arterial tonometry (EndoPat)

SECONDARY OUTCOMES:
Augmentation index | Baseline to 12 Weeks
  Arterial stiffness assessed as augmentation index using an automated blood pressure monitor (SphygmoCor)
Pulse wave velocity | Baseline to 12 Weeks
  Arterial stiffness assessed as carotid-femoral pulse wave velocity using an automated blood pressure monitor (SphygmoCor)
Endothelial cell protein expression | Baseline to 12 Weeks
  Protein expression will be assessed as an exploratory analysis for markers of nitric oxide bioavailability, inflammation, and/or oxidative stress will be measured by quantitative immunofluorescence in biopsied venous endothelial cells
Hemoglobin A1c | Baseline to 12 Weeks
  Blood hemoglobin A1C will be measured
Lipid profile | Baseline to 12 Weeks
  Blood lipid profiles will be measured
Nitric oxide metabolites | Baseline to 12 Weeks
  Blood nitrate/nitrite will be measured
ICAM-1 | Baseline to 12 Weeks
  Blood ICAM-1 will be measured
VCAM-1 | Baseline to 12 Weeks
  Blood VCAM-1 will be measured
Blood pressure | Baseline to 12 Weeks
  Brachial and Aortic blood pressure (systolic blood pressure, diastolic blood pressure, pulse pressure, aortic pressure) assessed using an automated blood pressure monitor (SphygmoCor)
Gut microbiota | Baseline to 12 Weeks
  Determine the effects on stool sample microbial populations
Plasma blueberry polyphenol metabolites | Baseline to 12 Weeks
  Targeted analysis of plasma metabolites by GC-MS and LC-MS

CONTACTS AND LOCATIONS:
Locations (1):
- Food and Nutrition Clinical Research Laboratory, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson SA, Figueroa A, Navaei N, Wong A, Kalfon R, Ormsbee LT, Feresin RG, Elam ML, Hooshmand S, Payton ME, Arjmandi BH. Daily blueberry consumption improves blood pressure and arterial stiffness in postmenopausal women with pre- and stage 1-hypertension: a randomized, double-blind, placebo-controlled clinical trial. J Acad Nutr Diet. 2015 Mar;115(3):369-377. doi: 10.1016/j.jand.2014.11.001. Epub 2015 Jan 8. PMID 25578927